CLINICAL TRIAL: NCT05143294
Title: Conectar Jugando: Effectiveness of a Modern Board Gamebased Cognitive Training to Improve Executive Function in Elementary Classrooms (6-12 Years Old) by a Cluster Controlled Trial
Brief Title: Conectar Jugando: Board Games in Elementary Classrooms (6-12 Years Old) to Improve Executive Functions
Acronym: CJ-Aula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brain In Game scientific-technical service (Other)
Collaborators: Atención, Familia, Infancia, Mayores (AFIM21) (Unknown); Mercurio Distribuciones (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NCT2021CJA
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Cognitive Change; Child Development
Keywords: executive function; modern board games; cognitive training; school-age children

STUDY DESIGN:
Intervention Model Description: Cluster RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modern board and card games group (Experimental): The program consisted of 12 one-hour intervention sessions. The sessions were biweekly with a total duration of 6 weeks. The modern board and card games used in the program were Bee Alert (Knizia, 2012), Monster Match (Gruhl & Weir, 2018), Kaleidos Junior (Albertarelli, 1997), Sherlock Express (Kermarrec, 2019), Alles Kanone! (Knizia, 2007), Halli Galli (Shafir, 1990), Bananazul (Warsch, 2019), Blurble (Bernard, 2013), La Morada Maldita (Ortiz, 2020), Dice Academy (Gobert, 2019) and Streams (Itsubaki, 2011). Play sessions will be held in subgroups of 3-5 children within the class group. In each session, each subgroup will play two games. The games used in the program have an average duration of approximately 20-30 minutes (filler games). All subgroups will play all games in the program the same number of times with the same rules. The game program will be the same in all participating centers to guarantee the homogeneity of its implementation.
  Interventions: Behavioral: Conectar Jugando Classroom Program
- Wait-list group (No Intervention): Wait-list. They will do the usual classes without modern board games. At the end of the post-intervention evaluation, the Conectar Jugando game program will be implemented under the same conditions as the experimental group.

INTERVENTIONS:
Behavioral: Conectar Jugando Classroom Program — Modern Board Games Intervention in Elementary Classrooms
  Arms: Modern board and card games group

SUMMARY:
Executive functions are cognitive processes that have been frequently related to adequate academic performance in the scientific literature. Current research aimed at training executive functions has found promising results using the modern board game as a cognitive tool in children. Considering the growing interest of teachers in this playful and possibly educational and cognitive resource, a game program for cognitive purposes has been designed to be used in primary classrooms. The main objective of the present study is to test the efficacy of a cognitive training program in the classroom based on modern board games in primary school students from ordinary schools (6 to 12 years old). For this, there will be an experimental group that will carry out the game program "Conectar Jugando" in the classroom implemented by the teachers of the participating centers, and a control group that will be on standby and will be compensated by carrying out the game program at the finalize the post-intervention evaluation. The classes of each school stage will be randomly assigned to an experimental group and a passive control group in each of the participating schools.

DETAILED DESCRIPTION:
As hypotheses, it is established that: i) the experimental group will present a significantly greater improvement in the neuropsychological tasks that measure executive functions compared to the passive control group after the intervention; ii) the experimental group will present a significantly greater improvement in the tests evaluated by their parents / teachers after the intervention compared to the passive control group; iii) the experimental group will present a significantly greater improvement in academic tests after the intervention compared to the passive control group. All hypotheses will be controlled for age, estimate of IQ and socioeconomic status, as well as previous experience in board games and other cognitive activities.

ELIGIBILITY:
Inclusion Criteria:

* be enrolled in an ordinary educational center, whether public, private or subsidized
* provide informed consent from both parents and the participant's agreement to participate in the study

Exclusion Criteria:

* comprehension difficulties due to language reasons
* sensory difficulties that make it impossible to carry out the program activities

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Visuospatial keep track task (Tamnes et al., 2010) | Baseline and post intervention (after 6 weeks)
  Change in visuospatial updating from baseline to post intervention. It consists of 9 trials of increasing difficulty in which colored faces move across the screen and it is necessary to remember the last position of each one.
Inhibition - Child Fish Flanker Task (Benzing et al., 2018) | Baseline and Post-intervention (after 6 weeks)
  Change in inhibition from baseline to post intervention. It is an adaptation of the classic Flanker Task in which fish must be fed by pressing the key that indicates the direction of the central fish. The inhibition measure is obtained by subtracting the reaction time of the pure block of congruent tests (5 fish going in the same direction) from the standard block that includes congruent and incongruent tests (the 4 fish that accompany the central fish can go in the same direction or the opposite).
Shifting - Child Fish Flanker Task (Benzing et al., 2018) | Baseline and Post-intervention (after 6 weeks)
  Change in shifting from baseline to post intervention. To obtain this measure, a mixed block is included in the fish flanker task in which trials of yellow fish and trials of red fish appear. When the fish are red, the central fish should be fed. When the fish are yellow, the fish from the sides should be fed. For both conditions, congruent and incongruent tests are presented. The subtraction of the reaction time from the standard block (only congruent and incongruent reds) to the mixed block (reds and yellows) gives rise to the shifting measure.
PREDISCAL (Pina-Paredes et al., 2020) | Baseline and Post-intervention (after 6 weeks)
  Change in academic competences from baseline to post intervention. Screening test that assesses Reading Fluency, Mathematical Fluency and Calculus in three timed written tasks.

SECONDARY OUTCOMES:
ATENTO - Family (Luque & Sánchez-Sánchez, 2019) | Baseline and Post-intervention (after 6 weeks)
  Change in behavioral executive functions from baseline to post intervention

OTHER OUTCOMES:
Reasoning - TONI-4 (Ruíz-Fernández, 2019) | Baseline
  It is a reasoning test in which series and matrices are presented that the child must complete with the available options so that the set makes sense. This measure will be used as a control variable.
Hollingshead Index (Hollingshead, 1975) | Baseline
  Sociodemographic data (age, sex, school year and socioeconomic status)
The Parent Play Beliefs Scale (PPBS) (Fogle & Mendez, 2006) | Baseline and Post-intervention (after 6 weeks)
  It consists of 30 items with 5 response options ranging from 1 (Disagree) to 5 (Strongly agree). Two subscales have been considered: a) Play support; b) Acedemic focus. The Play Support subscale refers to parents' positive beliefs about the relevance of play for children's development and about their participation in play with children. High scores on this subscale indicate that parents enjoy play, prioritize play, and view it as a means of teaching. The Academic focus subscale is made up of elements about the parents' emphasis on academic skills and the belief that play can promote their development. The Academic focus subscale is made up of elements about the parents' emphasis on academic skills and the belief that play can promote their development. High scores on this subscale would indicate that parents see the academic role of play as important.
Parent Survey of Typical Child Time Spent in Less-structured Activities (adapted from Barker et al., 2014) | Baseline
  In this survey, parents are asked (with the help of their children) about the time their children dedicate to less-structured and recreational activities using a using a 7-point scale (from lowest to highest frequency). High scores on each item mean a higher frequency in that activity. The sum of all the scores on each item (where 1= 'Never' and 7 = 'Daily') results in a typical less-structured activity score.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Education, Psychology and Social Work; University of Lleida, Lleida, Spain

REFERENCES:
- [Background] Barker JE, Semenov AD, Michaelson L, Provan LS, Snyder HR, Munakata Y. Less-structured time in children's daily lives predicts self-directed executive functioning. Front Psychol. 2014 Jun 17;5:593. doi: 10.3389/fpsyg.2014.00593. eCollection 2014. PMID 25071617
- [Background] Benzing V, Schmidt M, Jager K, Egger F, Conzelmann A, Roebers CM. A classroom intervention to improve executive functions in late primary school children: Too 'old' for improvements? Br J Educ Psychol. 2019 Jun;89(2):225-238. doi: 10.1111/bjep.12232. Epub 2018 Jun 26. PMID 29947142
- [Background] Tamnes CK, Ostby Y, Walhovd KB, Westlye LT, Due-Tonnessen P, Fjell AM. Neuroanatomical correlates of executive functions in children and adolescents: a magnetic resonance imaging (MRI) study of cortical thickness. Neuropsychologia. 2010 Jul;48(9):2496-508. doi: 10.1016/j.neuropsychologia.2010.04.024. Epub 2010 Apr 29. PMID 20434470